CLINICAL TRIAL: NCT02476942
Title: A Multicenter, Non-Interventional Study Evaluating Bleeding Incidence, Health-Related Quality of Life, and Safety in Patients With Hemophilia A Under Standard-of-Care Treatment
Brief Title: A Prospective Study to Collect High-Quality Documentation of Bleeds, Health-Related Quality of Life (HRQoL), and Safety Outcomes in Patients With Hemophilia A Treated With Standard-of-Care Treatment
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BH29768
Record Dates: First submitted 2015-06-03; First posted 2015-06-22 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Cohort A: Adults and Adolescents with FVIII Inhibitors: Adults and adolescents with hemophilia A of any severity with the presence of FVIII inhibitors will be observed.
  Interventions: Drug: Bypassing Agents
- Cohort B: Children with FVIII Inhibitors: Children with hemophilia A of any severity with the presence of FVIII inhibitors will be observed.
- Cohort C: Adults and Adolescents without FVIII Inhibitors: Adults and adolescents with severe hemophilia A without the presence of FVIII inhibitors will be observed.
  Interventions: Drug: FVIII Replacement

INTERVENTIONS:
Drug: Bypassing Agents — Episodic or prophylactic treatment with the use of bypassing agents must be documented for at least the last 6 months prior to the study. During the study, treatment for bleeds will be documented. The choice of coagulation product is at the discretion of the investigator according to local practice standards in this non-interventional study and there are no specific protocol-defined interventions.
  Groups: Cohort A: Adults and Adolescents with FVIII Inhibitors
Drug: FVIII Replacement — Episodic or prophylactic treatment with the use of FVIII replacement must be documented for at least the last 6 months prior to the study. During the study, treatment for bleeds will be documented. The choice of coagulation product is at the discretion of the investigator according to local practice standards in this non-interventional study and there are no specific protocol-defined interventions.
  Groups: Cohort C: Adults and Adolescents without FVIII Inhibitors

SUMMARY:
This non-interventional study will prospectively collect detailed, high-quality documentation of bleeds, HRQoL, and safety in patients with hemophilia A with or without FVIII inhibitors treated according to local routine clinical practice (receiving FVIII replacement or bypassing agents as either episodic or prophylactic treatment). Actual patients will be enrolled from routine clinical practice in this observational study.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: Patients greater than or equal to (>/=) 12 years of age at time of informed consent
* Cohort A: Diagnosis of congenital hemophilia A of any severity and documented history of high-titer inhibitor (that is, >/= 5 Bethesda units [BU])
* Cohort B: Pediatric patients less than (<) 12 years of age
* Cohort B: Diagnosis of congenital hemophilia A of any severity and documented history of high-titer inhibitor (that is, >/=5 BU)
* Cohort C: Patients >/=12 years of age
* Cohort C: Diagnosis of congenital hemophilia A and FVIII activity <1 percent (%)
* Cohort C: No prior history of a positive inhibitor against FVIII

Exclusion Criteria:

* Prior RO5534262 (not applicable if patient agrees that prior RO5534262 will preclude participation in a future investigational RO5534262 study)
* Bleeding disorder other than congenital hemophilia A
* Ongoing (or planned during the study) immune tolerance induction therapy with FVIII or FVIII prophylaxis if currently/previously exposed to an inhibitor
* Previous or concomitant thromboembolic disease
* Known human immunodeficiency virus (HIV) infection with cluster of differentiation (CD) 4 count <200 cells per microliter (cells/mcL)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia A with or without inhibitors against FVIII under standard-of-care treatment are to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Bleeds | Approximately 6 months (from Baseline until study completion)

SECONDARY OUTCOMES:
European Quality of Life-5 Dimensions (EQ-5D-5L) Questionnaire Score Among Adult and Adolescent Patients | Approximately 6 months (every 4 weeks from Baseline until study completion and on days that bleeds are reported)
Hemophilia A-Specific Quality of Life (Haem-A-QoL) Questionnaire Score Among Adult Patients | Approximately 6 months (every 4 weeks from Baseline until study completion)
Hemophilia-Specific Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Score | Approximately 6 months (every 4 weeks from Baseline until study completion)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (35):
- United States (10):
  - Santa Monica Oncology Center, Santa Monica, California
  - University of Colorado Denver, Children's Hospital, Aurora, Colorado
  - Georgetown Uni Medical Center; Lombardi Cancer Center, Washington D.C., District of Columbia
  - Winship Cancer Institute, Atlanta, Georgia
  - Tulane Uni Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital of Michigan; Pediatrics, Detroit, Michigan
  - Cornell Univ Medical College; Hematology-Oncolog, New York, New York
  - Oregon Health & Science Uni ; Dept of Pediatrics, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Bloodworks Northwest (formerly Puget Sound Blood Center); Hemophilia, Seattle, Washington
- Australia (2):
  - Royal Prince Alfred Hospital; Haematology, Camperdown, New South Wales
  - The Alfred Hospital, Melbourne; Thrombosis and Haemostasis Unit, Melbourne, Victoria
- China (3):
  - Peking Union Medical College Hospital, Beijing
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Tianjin Institute of Hematology & Blood Diseases Hospital, Tianjin
- ICIC, San José, Costa Rica
- Universitätsklinikum Bonn (AöR); Inst. für Experimentelle Hämatologie u. Transfusionsmedizin (IHT), Bonn, Germany
- Italy (2):
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico; Centro Emofilia e Trombosi "Angelo Bianchi e Bonomi", Milan, Lombardy
  - AOU Careggi; SOD Malattie Emorragiche, Florence, Tuscany
- Japan (6):
  - Nagoya University Hospital, Aichi
  - Hyogo College of Medicine Hospital, Hyōgo
  - St. Marianna University School of Medicine Hospital, Kanagawa
  - Hospital of the University of Occupational and Environmental Health,Japan, Kitakyushu-shi
  - Nara Medical University Hospital, Nara
  - Tokyo Medical University Hospital, Tokyo
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne; Klinika Hematologii i Transplantologii, Gdansk
  - SPSK Nr1 Klinika Hematoo&Transpl.Szpiku, Lublin
  - ALVAMED Lekarskie Gabinety Specjalistyczne, Poznan
  - Instytut Hematologii i Transfuzjologii; Klinika Zaburzeń Hemostazy i Chorób Wewnętrznych, Warsaw
- Charlotte Maxeke Johannesburg Hospital; Haemophilia Comprehensive Care Center, Johannesburg, South Africa
- Severance Hospital, Seoul, South Korea
- Spain (3):
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
  - Hospital Universitario la Fe; Servicio de Hematologia, Valencia
- National Taiwan Uni Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Oldenburg J, Shima M, Kruse-Jarres R, Santagostino E, Mahlangu J, Lehle M, Selak Bienz N, Chebon S, Asikanius E, Trask P, Mancuso ME, Jimenez-Yuste V, von Mackensen S, Levy GG. Outcomes in children with hemophilia A with inhibitors: Results from a noninterventional study. Pediatr Blood Cancer. 2020 Oct;67(10):e28474. doi: 10.1002/pbc.28474. Epub 2020 Aug 9. PMID 32776489